CLINICAL TRIAL: NCT03295591
Title: Optimizing the Selection of Patients With Metastatic Colorectal Cancer for Liver Resection - An Immuno-clinical Scoring System Incorporating Circulating Tumor Cell Enumeration and Clinical Factors
Brief Title: Circulating Tumor Cells in mCRC for Liver Resection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Lam Ka On, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: UW17-008
Record Dates: First submitted 2017-09-19; First posted 2017-09-28 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Metastatic Colorectal Cancer; Circulating Tumor Cell
Keywords: Metastatic colorectal cancer; Liver resection; Circulating tumor cells
MeSH Terms: conditions — Colorectal Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood in Streck tube will be processed for isolating circulating tumor cells and its DNA content for subsequent sequencing if feasible
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Diagnostic Test: Circulating tumor cell — Circulating tumor cell enumeration and sequencing

SUMMARY:
Resection of liver metastasis is potentially curative in patients with colorectal cancer bearing liver metastasis. However, early recurrence occurs in up to 30% in 3 months after liver resection. To optimize patient selection, the investigators propose to evaluate the the value of incorporating circulating tumor cells enumeration to clinical factors in a prospective study

DETAILED DESCRIPTION:
This is a single-center prospective study to evaluate the predictive value of circulating tumor cells (CTC) in patients with metastatic colorectal cancer who are planned to have curative resection of liver metastasis. Blood will be taken from patients within 7 days before liver resection. CTC enumeration is done by a highly-sensitive microfluidic platform for which CTC can be subsequently enumerated with or without sequencing performed. Patients are then followed up regularly with contrast CT scan for recurrence. The primary study endpoint is to define the cutoff value of CTC count in patients with early relapse < 6months after liver resection. Seventy-seven patients will be recruited in 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age>=18 years
2. Signed informed consent
3. Histologically or cytologically confirmed colorectal adenocarcinoma
4. Both primary tumor and liver metastases are amenable to curative resection.

Exclusion Criteria:

1. Presence of extrahepatic metastasis
2. History of other malignancies in the last 5 years
3. Patients unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with colorectal cancer and liver metastasis who are planned for liver resection
Sampling Method: Non-Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Cutoff value of CTC counts | Progression free survival at 6 months
  to identify patients with early relapse (<6 months) after liver resection as determined by the AUC under the ROC curve

SECONDARY OUTCOMES:
A immuno-clinical scoring system | Progression free survival at 6 months
  A system combining CTC count with clinical factors to stratify patients before liver resection
Progression free survival | up to 5 years
  Time from liver resection to date of relapse or date of death, whichever is earlier
Overall survival | up to 5 years
  Time from liver resection to date of death

CONTACTS AND LOCATIONS:
Overall Officials: Ka On Lam, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided